CLINICAL TRIAL: NCT01263951
Title: A Phase II Study of Everolimus and Sorafenib in Patients With Metastatic Differentiated Thyroid Cancer Who Have Progressed on Sorafenib Alone
Brief Title: Study of Everolimus and Sorafenib in Patients With Advanced Thyroid Cancer Who Progressed on Sorafenib Alone
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bayer (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19309; 812004 (Other: University of Pennsylvania IRB #1)
Record Dates: First submitted 2010-11-29; First posted 2010-12-21 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Differentiated metastatic thyroid cancer
MeSH Terms: interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus and sorafenib (Experimental): All patients will receive everolimus and sorafenib daily.
  Interventions: Drug: Everolimus; Drug: Sorafenib

INTERVENTIONS:
Drug: Everolimus — One 5 mg. tablet daily.
  Other Names: Afinitor
Drug: Sorafenib — 200 mg. twice daily.
  Other Names: Nexavar

SUMMARY:
The goal of this study is to determine the effect of combining everolimus and sorafenib in patients with metastatic differentiated thyroid cancer who progressed on sorafenib alone.

DETAILED DESCRIPTION:
The purpose of this research study is to:

1. Find out if sorafenib and everolimus prevent the growth of tumors that have grown when treated with sorafenib alone
2. Find out how long one might benefit from treatment with sorafenib and everolimus
3. Find out what side effects this drug may cause
4. Measure the amount of sorafenib and everolimus in the blood and see if "markers" can be found to help understand who might benefit from sorafenib and everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thyroid cancer, that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* All patients will have been required to have had sorafenib for entry and have had documented progression while on previous treatment with sorafenib.
* Measurable disease defined as at least one malignant lesion that can be accurately measured on computerized tomography (CT) and/or magnetic resonance imaging (MRI) scan.
* ECOG performance status < 2.
* Life expectancy greater than 3 months.
* Intellectual, emotional, and physical ability to comply with oral medication.

Exclusion Criteria:

* Restrictions regarding certain prior treatments will apply.
* Significant medical disease including: uncontrolled congestive heart failure; active symptoms of coronary artery disease, uncontrolled seizure disorder; active infection; uncontrolled diabetes mellitus; requirement for chronic high dose corticosteroid treatment (Topical or inhaled corticosteroids are allowed); requirement for concurrent immunosuppressive drug(s); active autoimmune disease.
* Organ allografts.
* Known HIV-infection (HIV testing is not required for participation).
* Pregnant or breast feeding. Women of childbearing potential and sexually active males must be advised to take precautions to prevent pregnancy during treatment
* History of second cancer (except adequately treated basal cell or squamous cell skin cancer, in situ treated cervical cancer, colon cancer or melanoma, or any other cancer for which the patient has been disease-free for three or more years).
* Known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
* Use of any experimental therapy within 4 weeks prior to baseline evaluations done prior to enrollment (with the exception of sorafenib which may be continued until treatment start). Therefore, all experimental treatments other than sorafenib must be discontinued 4 weeks prior to baseline studies or enrollment.
* Patients who did not previously tolerate sorafenib at 200 mg once daily are excluded from the study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-11; Primary Completion 2021-02-01 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of everolimus and sorafenib (progression free survival, objective response rate and stable disease) in patients with advanced differentiated thyroid cancer who have progressed on sorafenib alone. | Every 4 weeks

SECONDARY OUTCOMES:
To evaluate the secondary endpoints of best response in patients receiving everolimus and sorafenib. | Every 4 weeks
To perform correlative scientific studies to determine the relationship between clinical response to everolimus and sorafenib and multiple parameters including the mutational status of BRAF, N-RAS and other relevant cancer genes in the tumor. | Every 4 weeks
To investigate the effectiveness of mTOR and Raf kinase inhibition in surrogate tissue and tumor samples. | Every 4 weeks
To evaluate the activity of additional signaling pathways in surrogate tissue and tumor samples and explore their relevance to outcome measures. | Every 4 weeks
To evaluate the secondary endpoints of time to disease progression in patients receiving everolimus and sorafenib. | Every 4 weeks
To evaluate the secondary endpoints of duration of response in patients receiving everolimus and sorafenib. | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Brose, MD, PhD, Principal Investigator — Hospital of the University of Pennsylvania- Abramson Cancer Center
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not at this time